CLINICAL TRIAL: NCT02148770
Title: Modulating Functional Connectivity Between Eating-related Brain Areas by Neurofeedback
Brief Title: The Effect of Neurofeedback on Eating Behaviour
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 646/2013BO2
Record Dates: First submitted 2014-05-14; First posted 2014-05-28 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2015-06

CONDITIONS: Obesity; Eating Behaviour
Keywords: rt-fmri; self-control; eating behaviour; overweight; neurofeedback
MeSH Terms: conditions — Obesity; Feeding Behavior; Self-Control; Overweight | interventions — Neurofeedback

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurofeedback (Experimental): Neurofeedback training: Up-regulation of DLPFC.
  Interventions: Device: Neurofeedback
- Neurofeedback SHAM (Sham Comparator): Neurofeedback training: Sham-regulation of DLPFC.
  Interventions: Device: Neurofeedback

INTERVENTIONS:
Device: Neurofeedback — Networks involved in eating behaviour can be modified by neurofeedback training. We will perform a neurofeedback task using the technology of fMRI-based Brain Computer Interface (BCI). BCI approaches based on real-time fMRI (rtfMRI) allow voluntary regulation of brain regions. For the rtfMRI, a well-established setup will be used which translates the blood oxygen level dependent (BOLD) signal of a specific brain region of interest into a visual signal (e.g. moving bar) in real time using brain voyager® and matlab. The study will include 1 training-sessions In the up-regulation condition subjects will learn to up regulate their dlPFC. In the sham-condition subjects are get the same instructions, however they will receive sham feedback.
  Other Names: fMRI-based Brain Computer Interface (BCI); Neurofeedback training; rtfMRI

SUMMARY:
Neuroimaging is becoming increasingly common to investigate the neural networks underlying eating behaviour and food preference in normal-weight and obese humans. It has been observed that obese in comparison to lean individuals display altered activation patterns in networks of brain areas involved in reward, emotion and cognitive control. Interestingly, obese individuals who are capable of losing weight appear to have a stronger connectivity between areas related to food value and to the control of eating behaviour. The same areas are also associated with healthy food choices. It has been suggested that activation in the prefrontal control areas indirectly modulate valuation-related activity. Based on this, brain-related intervention strategies to support weight loss and long-lasting weight maintenance are of particular interest. Hence, we first want to examine the effect on eating behaviour of neurofeedback training-induced up-regulation of functional connectivity between reward- and impulse-related brain areas as a pilot, and second we want to examine up-regulation of the activity of prefrontal control brain areas.

DETAILED DESCRIPTION:
Primary objective: We want to investigate whether the training-induced up-regulation of the dorsal prefrontal cortex inhibits eating behaviour.

Study design: A parallel design. Half of the participants will learn to up-regulate activity of the dorsolateral prefrontal cortex (dlPFC), while the other participants will participate in sham-training sessions. Adherence to experimental conditions will be assigned randomly, based on the participants' enrolment in the study, balanced by gender and binge eating classification.

Study population: 50 overweight and obese (BMI 25-40 kg/m2), but otherwise healthy individuals, 18-65 years old.

Intervention: All participants will participate in a screening day, followed by one neurofeedback session day and a follow-up day. During the neurofeedback session, participants will undergo a 45 min real-time-fMRI-brain-computer-interface scan in order to learn to up-regulate dlPFC activation.

Main study parameters/endpoints:

1. The ability to up-regulate dlPFC activity.
2. Respective effects on eating behaviour. Nature and extent of the burden and risks associated with participation: Participants will be scanned once (fMRI). Functional MRI is a safe and non-invasive technique.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects
* Age 18-65 years at start of the study
* Body Mass Index (BMI) between 25 and 40 kg/m2
* Informed consent to study protocol
* Willingness to be informed about chance findings of pathology and approval of the disclosure of this information to the general physician (see Informed Consent)
* Fulfilment of the criteria for blood donors according to the "Richtlinien zur Gewinnung von Blut und Blutbestandteilen und zur Anwendung von Blutprodukten", in particular Hb ≥ 135 g/l (8,37 mmol/l; Bundesärztekammer 2010)

Exclusion Criteria:

* Subjects who have a non-removable metal object in or at their body, such as, for ex-ample:

  * Heart pace-maker
  * Artificial heart valve
  * Metal prosthesis
  * Metallic implants (screws, plates from operations, etc.)
  * Metal splinters / grenade fragments
  * Non-removable dental braces
  * Acupuncture needles
  * Insulin pump
  * Intraport, etc.
  * In field strengths of over 1.0 T also: tattoos, eye lid-shadow
* Current weight loss regimens
* Limited temperature perception and/or increased sensitivity to warming of the body
* Pathological hearing ability or an increased sensitivity to loud noises
* Claustrophobia
* Lack of ability to give informed consent
* Operation less than three month ago
* Simultaneous participation in other studies
* Acute illness or infection during the last 4 weeks
* Neurological disorder or injury
* Moderate or severe head injury
* Severe psychotic illness
* Intake of antidepressants / antipsychotics
* Participation in other studies with blood withdrawals or blood donation in previous and subsequent 2 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-11; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Activity in the dlPFC during the training-session | 1 day
  Differences in dlPFC activity between baseline and after up-regulation during the neurofeedback training session, as well as the difference between the treatment and the sham groups (ANCOVA approach).

SECONDARY OUTCOMES:
Food intake | 4 weeks
  Snack consumption during the snack test, comparing pre vs post neurofeedback session, and between the two groups (ANCOVA approach).
Preferred food (healthy or unhealthy food). | 4 weeks
  Differences in food choice (healthy vs unhealthy) pre compared to post neurofeedback session and between the two groups (ANCOVA approach).
Weight | 4 weeks
  Difference in weight before and after training

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Hallschmid, PhD, Principal Investigator — University Tuebingen
Locations (1):
- UKT and MPI, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
We will share the data inside the EU-consortium

REFERENCES:
- [Background] Weiskopf N, Scharnowski F, Veit R, Goebel R, Birbaumer N, Mathiak K. Self-regulation of local brain activity using real-time functional magnetic resonance imaging (fMRI). J Physiol Paris. 2004 Jul-Nov;98(4-6):357-73. doi: 10.1016/j.jphysparis.2005.09.019. Epub 2005 Nov 10. PMID 16289548
- [Background] Sitaram R, Caria A, Veit R, Gaber T, Rota G, Kuebler A, Birbaumer N. FMRI brain-computer interface: a tool for neuroscientific research and treatment. Comput Intell Neurosci. 2007;2007:25487. doi: 10.1155/2007/25487. PMID 18274615
- [Derived] Spetter MS, Malekshahi R, Birbaumer N, Luhrs M, van der Veer AH, Scheffler K, Spuckti S, Preissl H, Veit R, Hallschmid M. Volitional regulation of brain responses to food stimuli in overweight and obese subjects: A real-time fMRI feedback study. Appetite. 2017 May 1;112:188-195. doi: 10.1016/j.appet.2017.01.032. Epub 2017 Jan 25. PMID 28131758
- See also: Overview of main EU-project. — http://www.braintrainproject.eu/